CLINICAL TRIAL: NCT05638711
Title: Built-in Calculator Optimizes Continuous Veno-venous Hemofiltration Prescription and Improves Therapeutic Quality in Critically-ill Acute Kidney Injury Patients
Status: Completed | Type: Observational
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: haomingwu
Record Dates: First submitted 2022-11-15; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: CVVH; Filtration Fraction; Built-in Culculator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before group: * Patient: ICU patients received CVVH between 2019/01/01 - 2020/10/01 (before utilization of built-in calculator)
  * received regular protocol of ICU patient care (same in two groups)
- After group: * Patient: ICU patients received CVVH between 2020/10/01 - 2021/12/31 (after utilization of built-in calculator)
  * received regular protocol of ICU patient care (same in two groups)
  Interventions: Device: Built-in calculator to calculate Filtration fraction

INTERVENTIONS:
Device: Built-in calculator to calculate Filtration fraction — A calculator built in electronic CVVH prescription system to calculate Filtration fraction
  Groups: After group

SUMMARY:
The goal of this observational study is to compare in ICU patients received CVVH treatment. The main questions it aims to answer are:

Control of Filtration fraction by built-in calculator

* Reduced filter clotting and prolong filter lifespan
* Improve patient mortality Participants will divided into before group and after group based on the day when built-in calculator for calculating Filtration fraction was utilized.

Researchers will compare before group to see if there were differences in clotting events, filter downtime, filter lifespan, mortality, etc.

DETAILED DESCRIPTION:
# built-in calculator for calculating Filtration fraction

* The calculator was built in prescription system since 2020/10/01
* providing tempt filtration fraction for operators to adjust CVVH dose
* the protocol of patient care didn't change between before and after group.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients received CVVH during 2019~2021 (3 years) in our hospital

Exclusion Criteria:

* under age of 20, pregnant, or with HIV infection

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients received CVVH during 2019~2021 (3 years) in our hospital, and excluded patients under age of 20, pregnant, or with HIV infection
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days, 60 days, "through study completion, an average of 1.5 year" mortality in ICU and in Hospital
  Patient death

SECONDARY OUTCOMES:
Filter clotting events | "through the complete treatment course hours, an average of 24 hours"
  Filter clotting events
Filter lifespan | "through the complete treatment course hours, an average of 24 hours"
  average treatment time per filter
electrolytes_1 | the last record received before CVVH (in an average of 1 hour), the first record received CVVH after 24 hours, the first record received after CVVH (in an average of 1 hour)
electrolytes_2 | the last record received before CVVH (in an average of 1 hour), the first record received CVVH after 24 hours, the first record received after CVVH (in an average of 1 hour)
  K
electrolytes_3 | the last record received before CVVH (in an average of 1 hour), the first record received CVVH after 24 hours, the first record received after CVVH (in an average of 1 hour)
  Ca
electrolytes_4 | the last record received before CVVH (in an average of 1 hour), the first record received CVVH after 24 hours, the first record received after CVVH (in an average of 1 hour)
  P
acid-base balance_1 | the last record received before CVVH (in an average of 1 hour before CVVH treatment), the first record received CVVH after 24 hours (in an average of 1 hour after CVVH treatment), the first record received after CVVH (in an average of 1 hour after CVVH)
  pH
acid-base balance_2 | the last record received before CVVH (in an average of 1 hour before CVVH treatment), the first record received CVVH after 24 hours (in an average of 1 hour after CVVH treatment), the first record received after CVVH (in an average of 1 hour after CVVH)
  bicarbonate
Filter downtime | "through the complete treatment course hours, an average of 24 hours"
  downtime between filter replacement
others_1 | the last record received before CVVH (in an average of 1 hour before CVVH treatment), the first record received CVVH after 24 hours (in an average of 1 hour after CVVH treatment), the first record received after CVVH (in an average of 1 hour after CVVH)
  body temperature
others_2 | the last record received before CVVH (in an average of 1 hour before CVVH treatment), the first record received CVVH after 24 hours (in an average of 1 hour after CVVH treatment), the first record received after CVVH (in an average of 1 hour after CVVH)
  platelet

CONTACTS AND LOCATIONS:
Locations (1):
- Shuang-Ho Hospital, New Taipei City, Zhonghe District, Taiwan

IPD SHARING:
Plan to Share IPD: No
there is currently no plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Result] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Result] Davenport A. Continuous renal replacement therapies in patients with acute neurological injury. Semin Dial. 2009 Mar-Apr;22(2):165-8. doi: 10.1111/j.1525-139X.2008.00548.x. PMID 19426422
- [Result] Rabindranath K, Adams J, Macleod AM, Muirhead N. Intermittent versus continuous renal replacement therapy for acute renal failure in adults. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD003773. doi: 10.1002/14651858.CD003773.pub3. PMID 17636735
- [Result] Wang AY, Bellomo R. Renal replacement therapy in the ICU: intermittent hemodialysis, sustained low-efficiency dialysis or continuous renal replacement therapy? Curr Opin Crit Care. 2018 Dec;24(6):437-442. doi: 10.1097/MCC.0000000000000541. PMID 30247213
- [Result] Karkar A, Ronco C. Prescription of CRRT: a pathway to optimize therapy. Ann Intensive Care. 2020 Mar 6;10(1):32. doi: 10.1186/s13613-020-0648-y. PMID 32144519
- [Result] Tsujimoto Y, Fujii T. How to Prolong Filter Life During Continuous Renal Replacement Therapy? Crit Care. 2022 Mar 22;26(1):62. doi: 10.1186/s13054-022-03910-8. PMID 35337352
- [Result] Tsujimoto H, Tsujimoto Y, Nakata Y, Fujii T, Takahashi S, Akazawa M, Kataoka Y. Pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2020 Mar 13;3(3):CD012467. doi: 10.1002/14651858.CD012467.pub2. PMID 32164041
- [Result] Tsujimoto Y, Miki S, Shimada H, Tsujimoto H, Yasuda H, Kataoka Y, Fujii T. Non-pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2021 Sep 14;9(9):CD013330. doi: 10.1002/14651858.CD013330.pub2. PMID 34519356
- [Result] Joannidis M, Oudemans-van Straaten HM. Clinical review: Patency of the circuit in continuous renal replacement therapy. Crit Care. 2007;11(4):218. doi: 10.1186/cc5937. PMID 17634148
- [Result] Cottle D, Mousdale S, Waqar-Uddin H, Tully R, Taylor B. Calculating evidence-based renal replacement therapy - Introducing an excel-based calculator to improve prescribing and delivery in renal replacement therapy - A before and after study. J Intensive Care Soc. 2016 Feb;17(1):44-50. doi: 10.1177/1751143715603383. Epub 2015 Sep 21. PMID 28979457
- [Result] Griffin BR, Thomson A, Yoder M, Francis I, Ambruso S, Bregman A, Feller M, Johnson-Bortolotto S, King C, Bonnes D, Dufficy L, Wu C, Bansal A, Tad-Y D, Faubel S, Jalal D. Continuous Renal Replacement Therapy Dosing in Critically Ill Patients: A Quality Improvement Initiative. Am J Kidney Dis. 2019 Dec;74(6):727-735. doi: 10.1053/j.ajkd.2019.06.013. Epub 2019 Sep 17. PMID 31540789
- [Result] Ruiz EF, Ortiz-Soriano VM, Talbott M, Klein BA, Thompson Bastin ML, Mayer KP, Price EB, Dorfman R, Adams BN, Fryman L, Neyra JA; University of Kentucky CRRT Quality Assurance Group. Development, implementation and outcomes of a quality assurance system for the provision of continuous renal replacement therapy in the intensive care unit. Sci Rep. 2020 Nov 26;10(1):20616. doi: 10.1038/s41598-020-76785-w. PMID 33244053
- [Result] Honore PM, Spapen HD. What a Clinician Should Know About a Renal Replacement Membrane? J Transl Int Med. 2018 Jun 26;6(2):62-65. doi: 10.2478/jtim-2018-0016. eCollection 2018 Jun. No abstract available. PMID 29984198
- [Result] Yessayan L, Yee J, Frinak S, Szamosfalvi B. Continuous Renal Replacement Therapy for the Management of Acid-Base and Electrolyte Imbalances in Acute Kidney Injury. Adv Chronic Kidney Dis. 2016 May;23(3):203-10. doi: 10.1053/j.ackd.2016.02.005. PMID 27113697
- [Result] Kraut JA, Madias NE. Metabolic acidosis: pathophysiology, diagnosis and management. Nat Rev Nephrol. 2010 May;6(5):274-85. doi: 10.1038/nrneph.2010.33. Epub 2010 Mar 23. PMID 20308999
- [Result] Rocktaschel J, Morimatsu H, Uchino S, Ronco C, Bellomo R. Impact of continuous veno-venous hemofiltration on acid-base balance. Int J Artif Organs. 2003 Jan;26(1):19-25. doi: 10.1177/039139880302600104. PMID 12602465
- [Result] Leypoldt JK, Pietribiasi M, Echeverri J, Harenski K. Modeling acid-base balance during continuous kidney replacement therapy. J Clin Monit Comput. 2022 Feb;36(1):179-189. doi: 10.1007/s10877-020-00635-3. Epub 2021 Jan 3. PMID 33389356